CLINICAL TRIAL: NCT04843553
Title: Nicotinamide for Prevention of Pre-malignant Actinic Keratosis in Kidney Transplant Recipients: A Pilot Study
Brief Title: Nicotinamide for Prevention of Pre-malignant Actinic Keratosis in Kidney Transplant Recipients
Acronym: NICE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Rhode islandHospital
Record Dates: First submitted 2021-04-12; First posted 2021-04-13 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Actinic Keratoses
Keywords: Nicotinamide, AKs
MeSH Terms: conditions — Keratosis, Actinic | interventions — Niacinamide; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Research Pharmacists used list provided by biostatistician to fill unidentified (except for patient name) pill bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active (Active Comparator): Participants receiving oral vitamin B-3
  Interventions: Drug: Oral Nicotinamide
- placebo (Placebo Comparator): Participants receiving oral inactive pill
  Interventions: Drug: Oral Nicotinamide

INTERVENTIONS:
Drug: Oral Nicotinamide
  Other Names: Vitamin B-3

SUMMARY:
Skin cancers and pre-cancerous growths (called actinic keratoses, "AKs"), that aren't melanomas, develop in patients with a kidney transplant at excessive rates. When these pre-cancerous AKs, and "non-melanoma" skin cancers occur in kidney transplant patients, they tend to be aggressive, and require frequent medical procedures, often surgery, for the removal of the skin cancers. If not removed adequately the pre-cancers can develop into skin cancers, and the skin cancers, if not removed, may spread, and even cause death. Reducing the occurrence and complications of these skin cancers and pre-cancers in kidney transplant patients with a safe, effective, well-tolerated treatment taken by mouth would be an important medical advance.

We are testing oral nicotinamide (NAM)-a B-vitamin compound-for that purpose. Approximately fifty kidney transplant patients who have had at least one non-melanoma skin cancer in the past, will be given randomized to receive NAM, 1 gram twice daily by mouth, or identical pills without NAM, and followed for 1 year to see if NAM treatment reduces the numbers of pre-cancerous AKs, and non-melanoma skin cancers they develop. Patients will be asked to come to the clinic for 3 follow up visits (every 4 months for up to 12 months). They will receive a full body skin exam by a dermatologist, have detailed counting of AKs and biopsies for any suspicious lesions as standard of care. Blood will also be drawn as well as a urine sample obtained at each visit for safety assessment and storage. We will also ask them to answer a series of questions about dietary patterns and intake of whole foods and supplements.

DETAILED DESCRIPTION:
Non-melanoma cutaneous carcinomas [NMSCs], predominantly squamous cell carcinomas [SCCs], as well as basal cell carcinomas [BCCs], are the most common malignancies occurring in kidney transplant recipients [KTRs]. SCCs and BCCs, account for more than 90% of NMSCs in KTRs. New NMSCs in KTRs with a prior NMSC develop at 3-times the rate reported in non-KTRs with the same clinical history. The unique aggressiveness of SCCs in KTRs increases patient morbidity, due to the high rate of new lesions requiring treatment, frequently surgical excision. This non-fatal morbidity also results in significant medical costs. KTR SCCs have a greater potential for metastasis, and death. Reduction in the incidence and complications associated with SCCs, in particular, and more generally, overall NMSCs, as well as Actinic Keratoses, would mark a significant advance in the management of KTRs.

Specific Aims of this study are: To evaluate the effects of oral nicotinamide 2 grams/day, given in two divided doses, for 12-months, versus matched placebo, on the total number of actinic keratoses which develop in stable chronic kidney transplant recipients with a history of at least one non-melanoma skin cancer; To demonstrate our ability to create a system for diagnosing, capturing, and recording all new non-melanoma skin cancers which develop in stable chronic kidney transplant recipients with a history of at least one non-melanoma skin cancer while receiving oral nicotinamide 2 grams/day, given in two divided doses, for 12-months, versus matched placebo; To evaluate the effects of oral nicotinamide 2 grams/day, given in two divided doses, for 12-months, versus matched placebo, on sirtuin enzymatic activity in chronic kidney transplant recipients with a history of at least one non-melanoma skin cancer; To evaluate the safety and tolerability of oral nicotinamide 2 grams/day, given in two divided doses, for 12-months, versus matched placebo, in stable chronic kidney transplant recipients with a history of at least one non-melanoma skin cancer; To evaluate the effects of oral nicotinamide 2 grams/day, given in two divided doses, for 12-months, versus matched placebo, on serum phosphorus concentrations in stable chronic kidney transplant recipients with a history of at least one non-melanoma skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant ≥ 12-months ago
* ongoing, standard immunosuppression regimen
* current CKD
* EPI estimated (43)
* glomerular filtration rate (eGFR) ≥ 15 ml/min per 1.73 m2)
* Prior history of at least one NMSC

Exclusion Criteria:

* Kidney transplant <12-months ago, treatment for acute rejection <= 3-months ago, or current eGFR< 20
* Known history of active liver disease/ transaminitis [alanine aminotransferase, ALT > 1.5 X upper limit of normal]
* Serum phosphorus < 2.0 mg/dL or average ≤ 100 × 10(9)/mL platelets
* Internal malignancy, metastatic SCC, or invasive melanoma within the past 5-years
* Overwhelming numbers of current skin cancers or large areas of confluent skin cancer at baseline preventing accurate assessment and counting of new skin cancers
* Field treatment for AKs within the past 4-weeks, preventing accurate assessment of AKs
* Patients begun on acitretin or other oral retinoids, or mTOR inhibitors within the past 6-months (If stably taking for more than six months, they may participate)
* Gorlin's syndrome or other genetic skin cancer syndrome
* Patients unavailable for follow-up for the duration of the study because of social/ geographical reasons, or general frailty
* Pregnancy or lactation (all women of childbearing will be required to use contraception throughout the study)
* Patients taking supplemental NAM within the past 4-weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Effects of oral nicotinamide on AKs | 12 months
  To evaluate the effects of oral nicotinamide 1gram/day, given in two divided doses, for 9- 12-months, versus matched placebo, on the total number of actinic keratoses which develop in stable chronic kidney transplant recipients with a history of at least one non-melanoma skin cancer (keratinocyte carcinoma).
  To evaluate the effects of oral nicotinamide 1gram/day, given in two divided doses, for 9- 12-months, versus matched placebo, on the total number of actinic keratoses which develop in stable chronic kidney transplant recipients with a history of at least one non-melanoma skin cancer (keratinocyte carcinoma).

CONTACTS AND LOCATIONS:
Overall Officials: Reginald m Gohh, Principal Investigator — Rhode Island Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers HW, Weinstock MA, Feldman SR, Coldiron BM. Incidence Estimate of Nonmelanoma Skin Cancer (Keratinocyte Carcinomas) in the U.S. Population, 2012. JAMA Dermatol. 2015 Oct;151(10):1081-6. doi: 10.1001/jamadermatol.2015.1187. PMID 25928283
- [Background] Hartevelt MM, Bavinck JN, Kootte AM, Vermeer BJ, Vandenbroucke JP. Incidence of skin cancer after renal transplantation in The Netherlands. Transplantation. 1990 Mar;49(3):506-9. doi: 10.1097/00007890-199003000-00006. PMID 2316011
- [Background] Webb MC, Compton F, Andrews PA, Koffman CG. Skin tumours posttransplantation: a retrospective analysis of 28 years' experience at a single centre. Transplant Proc. 1997 Feb-Mar;29(1-2):828-30. doi: 10.1016/s0041-1345(96)00152-2. No abstract available. PMID 9123544